CLINICAL TRIAL: NCT06494423
Title: Supportive Care Intervention Development to Address Employment Concerns After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Employment Support After Hematopoietic Stem Cell Transplantation
Acronym: WorkS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kathleen Lyons, ScD, OTR/L, Professor, Occupational Therapy, MGH Institute of Health Professions
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024P000290
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Return to Work

STUDY DESIGN:
Intervention Model Description: A single arm proof-of-concept trial with up to 35 HSCT survivors reporting employment concerns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Work Support Intervention (Experimental): This is a single arm proof-of-concept trial with up to 35 HSCT recipients reporting employment concerns. We will refine and preliminarily evaluate a Work Support (WorkS) self-management intervention designed to catalyze return-to-work self-efficacy.
  Interventions: Behavioral: Work Support (WorkS)

INTERVENTIONS:
Behavioral: Work Support (WorkS) — The WorkS intervention entails two structured visits with a research team member initiated 6-months post-HSCT, which is the earliest point at which most HSCT survivors can safely consider returning to work. The sessions are focused on 1) identifying challenges of navigating work and illness; 2) linking survivors with psychological, rehabilitative, governmental, and community resources that can promote recovery and well-being; and 3) communicating with employers regarding the necessary work modifications to achieve mutual goals.

SUMMARY:
This is a feasibility study of a Work Support (WorkS) intervention designed to ameliorate employment challenges for people preparing to return to work after allogeneic stem cell transplantation. The aim of this study is to evaluate "proof of concept" by:

1. examining the feasibility and acceptability of the WorkS intervention and the study procedures, and
2. exploring the preliminary effects of WorkS for improving patient-reported return-to-work self-efficacy, work status, quality of life, and financial toxicity.

DETAILED DESCRIPTION:
Participants will be recruited from MGH Cancer Center. The intervention will be delivered at MGH Institute of Health Professions (IHP) and investigators at MGH IHP will be involved in recruiting participants and collecting/managing data.

Participants will be enrolled in the study for approximately six months following the schedule below:

* Enrollment into study: HSCT recipients will be recruited into the study approximately six months post HSCT (+/- one month).
* Baseline assessment: To be completed within 3 weeks of completing informed consent.
* WorkS Appointment #1 and #2: To be completed within a 2-month period after completing the baseline assessment. Ideally, the appointments will be approximately one month apart, but can be timed whenever in the 2-month window that is preferred by the participant.
* Exit assessment: To be completed within 3 weeks of completing Appointment 2.
* Final assessment: Return to work status at 12 months post HSCT (+/- three weeks)

ELIGIBILITY:
Inclusion Criteria:

* Received an allogeneic HSCT within the past six months to treat a hematological malignancy.
* Screen positive for work-related concerns (i.e., responds "yes" to the question, "Are you concerned about your ability to return to work in the coming six months?")

Exclusion Criteria:

* Patients with acute psychiatric or cognitive conditions which the treating clinician believes prohibits informed consent or compliance with the study procedures
* We will not enroll the following special populations: adults unable to consent, individuals not yet adults, pregnant women, and prisoners.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Screening Rate | At screening
  Number of patients screened / Number undergoing HSCT during study period
Eligibility Rate | At screening
  Number of patients screening positive & eligible / Number screened
Enrollment Rate | Up to 2 months
  Number of participants who attended the WorkS sessions / Number enrolled; Enrollment rate of at least 50% will indicate feasibility.
Intervention completion Rate | Up to 2 months
  Number of participants who attended the WorkS sessions / Number enrolled; Feasible if at least 80% of participants complete two sessions.
Assessment Completion Rate | Up to 6 months
  Number participants completing each of the three study assessments/ Number of participants enrolled

SECONDARY OUTCOMES:
Working Status | 6 months
  We will ask questions about the work status at the time of diagnosis, including the job title, average number of hours worked per week, the number of years at that worksite, the degree to which they get support from superiors at work, the flexibility of their workplace, the importance of and motivation for work, the degree to which their job is physically demanding, the degree to which their job is cognitively demanding, and the degree to which their job is psychologically demanding. We will also ask about the degree of certainty that the participant will return to the same job once they are cleared to return to work and the estimated timeframe for return to work.
Financial Toxicity | 2 months
  We will use the Functional Assessment of Chronic Illness Therapy-Comprehensive Score of Financial Toxicity (FACIT-COST) questionnaire to assess financial distress. The FACIT-COST is a 12-item patient-reported outcome measure that describes financial distress experienced by patients with cancer.
Quality of Life: Functional Assessment of Cancer Therapy - Bone Marrow Transplant | 2 months
  We will use the Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) scale to assess quality of life. The FACT-BMT is a 50-item, patient-reported measure that describes five dimensions of quality of life in bone marrow transplant patients: social well-being, physical well-being, functional well-being, emotional well-being and transplant-specific concerns.
Return to Work Self-Efficacy | 2 months
  The 11-item Return to Work Self-Efficacy Scale (RTWSE-11)[16] quantifies an individual's confidence in their ability to work fully and perform work tasks.
Concerns Regarding Work | 2 months
  We will ask the following open-ended question and record the response verbatim: "What concerns do you have about returning to work (either your previous job or if you seek or find a new job)?"
Utility of Intervention | 2 months
  Participants will rate their degree of agreement with statements regarding the utility of the workbook and the consultation. They will rate agreement on a five point scale where "1" is "strongly disagree" and "5" is "strongly agree."

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Lyons, ScD, OTR/L, Principal Investigator — MGH Institute of Health Professions
Locations (1):
- MGH Cancer Center, Boston, Massachusetts, United States